CLINICAL TRIAL: NCT01724827
Title: Ceramic Versus Composite in the Treatment by Inlays or Onlays of Posterior Teeth Affected by Tooth Substance Loss : a Multicenter Randomized Controlled Trial
Brief Title: Ceramic Versus Composite in the Treatment of Posterior Teeth by Inlays or Onlays
Acronym: CECOIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); Hôpital Charles Foix (Other); Hôtel Dieu - Service d'odontologie (Toulouse) (Unknown); Dental practitionners (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110129
Record Dates: First submitted 2012-09-10; First posted 2012-11-12 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Dental Caries; Inlays
Keywords: Dental caries; inlays; composite resins; IPS-Empress ceramic; bicuspid; FDI dental restorations evaluation criteria
MeSH Terms: conditions — Dental Caries; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ceramic (Active Comparator): Leucite-reinforced glass ceramic (Empress CAD, Ivoclar Vivadent)
  Interventions: Device: ceramic (Empress CAD, Ivoclar Vivadent)
- composite (Active Comparator): Nanohybrid composite resin (Lava Ultimate, 3M Espe)
  Interventions: Device: composite (Lava Ultimate, 3M Espe)

INTERVENTIONS:
Device: ceramic (Empress CAD, Ivoclar Vivadent) — Leucite-reinforced glass ceramic (Empress CAD, Ivoclar Vivadent)
  Arms: ceramic
Device: composite (Lava Ultimate, 3M Espe) — Nanohybrid composite resin (Lava Ultimate, 3M Espe)
  Arms: composite

SUMMARY:
The main purpose of this trial is to determine which material, between ceramic and composite, is best to manufacture dental inlays and onlays in the treatment of moderate dental substance losses, generally due to dental caries. Restorations will be done using direct Computer Assisted Design and Manufacturing (CAD-CAM). Another aim of this study is to determine which factors influence the success of these restorations.

DETAILED DESCRIPTION:
WHO estimates dental caries prevalence to be over 90% adults worldwide. When tooth substance loss due to the decayed tissue is small, a filling is done by the dentist directly. When the substance loss is important, dentists often treat it with a crown, which presents the disadvantage of further mutilating the tooth. An intermediate technique consists in manufacturing an inlay or an onlay: these restorations become more and more common since they are a minimally invasive solution in such cases. Inlays and onlays can be made of metal, ceramic or composite. Patients tend to refuse metallic restorations, so that dentists generally have to choose between composite and ceramic. Composite wears whereas ceramics fracture. Published in vitro studies provide possible answers to which material is most effective but very few clinical studies have been conducted to confirm them. Material\'s choice for inlay manufacturing is thus more country-based than evidence-based (Most french dentists choose composite while US dentists prefer ceramics for example). The main objective of this trial is to compare the clinical performance of ceramic and composite inlays/onlays. Other objectives include looking for the prognostic factors of these restorations and validating the criteria proposed by the World Dental Federation (FDI) to evaluate dental restorations.

ELIGIBILITY:
Inclusion criteria :

* patient aged 18-70,who tolerates restorative procedures and presents a moderate-sized dental caries or restoration (that needs to be replaced) necessitating an inlay/onlay restoration.

Exclusion criteria :

* allergy to one of the materials employed, bruxism, severe or acute periodontal or carious disease, poor oral hygiene
* Tooth presents a mobility > II, a periodontal socket > 3mm or supports a removable partial denture

Randomization criterium :

* tooth necessitates an inlay-onlay restoration after caries or former restoration removal

Exclusion from randomization criteria :

* subgingival margin after cavity preparation, rubber dam cannot be placed, all tooth cuspids need to be covered by the restoration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
FDI criteria for dental restorations assessment | at 2 years
  2 independent evaluators The primary outcome will consist in the FDI instrument for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010 . This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome.

SECONDARY OUTCOMES:
Restoration survival analysis | at 2 years
  The primary outcome will consist in the FDI instrument for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010 . This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome.
wear | at 2 years
  The primary outcome will consist in the FDI instrument for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010 . This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome.
overall quality of the restoration | at 2 years
  The primary outcome will consist in the FDI instrument for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010 . This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome.
FDI instrument validity data | at 2 years
  The primary outcome will consist in the FDI instrument for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010 . This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually.The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: hélène fron chabouis, DDS, MSc, Study Director — APHP, Hôpital Charles Foix, Service d'odontologie, Ivry-sur-Seine, France ; Faculté de chirurgie dentaire, Service de biomatériaux (URB2i EA4462), Université Paris Descartes, Sorbonne Paris Cité, Montrouge, France.
Locations (4):
- France (4):
  - Hôpital Charles Foix (APHP), Service d'odontologie, Ivry-sur-Seine
  - Dental pratice, Lyon
  - Dental pratice, Paris
  - Hôtel Dieu, Service d'odontologie, Toulouse

REFERENCES:
- [Result] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Science Committee Project 2/98--FDI World Dental Federation study design (Part I) and criteria for evaluation (Part II) of direct and indirect restorations including onlays and partial crowns. J Adhes Dent. 2007;9 Suppl 1:121-47. PMID 18341239
- [Result] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Derived] Fron Chabouis H, Prot C, Fonteneau C, Nasr K, Chabreron O, Cazier S, Moussally C, Gaucher A, Khabthani Ben Jaballah I, Boyer R, Leforestier JF, Caumont-Prim A, Chemla F, Maman L, Nabet C, Attal JP. Efficacy of composite versus ceramic inlays and onlays: study protocol for the CECOIA randomized controlled trial. Trials. 2013 Sep 3;14:278. doi: 10.1186/1745-6215-14-278. PMID 24004961
- See also: Cecoia website — http://www.cecoia.fr